CLINICAL TRIAL: NCT01846910
Title: Prepare to Quit - A Randomized Clinical Trial to Help People Quit Smoking in a Community Dental Clinic Setting
Brief Title: Prepare to Quit - A Clinical Trial to Help People Quit Smoking in a Community Dental Clinic Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Douglas James Brothwell, Associate Dean (Academic), University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2013:118
Record Dates: First submitted 2013-04-30; First posted 2013-05-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Smoking; Smoking Cessation
Keywords: Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Tooth Bleaching; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Counseling (Active Comparator): The extended counseling group will receive one to three, 45-minute individual motivational counseling sessions using a motivational interviewing approach to Express empathy, Develop discrepancy, Roll with resistance, and Support self-efficacy.
  Interventions: Behavioral: Motivational Counseling
- Tooth Whitening Incentive (Experimental): The tooth whitening group will receive all of the interventions previously described for the Motivational Counseling Group, and as an extra incentive against relapse, will also be offered complimentary tooth whitening procedures if biochemically verified as tobacco-free by Carbon Monoxide monitor (bleaching at 3-weeks, whitening strips at 3-months, and whitening touch-up at 1 year).
  Interventions: Behavioral: Tooth Whitening; Behavioral: Motivational Counseling

INTERVENTIONS:
Behavioral: Tooth Whitening — 1. A dental check-up will ensure the absence of contraindications to tooth whitening (cavities, soft tissue pathology, severe periodontitis) 2. Removal of calculus, plaque, or stains with a dental polishing 3. Treatment time is approximately 1 hour total4. Lips are retracted, tongue protector is placed and protective eyewear used 5. Saliva is suctioned and teeth are air dried 6. A liquid rubber dam material is applied to protect gums and cured by visible light. 7. The bleaching material is placed on the enamel surface of the involved teeth and is replaced if drying occurs 8. After 15 minutes, the bleach is suctioned, mouth rinsed and process repeated 9. Three to four applications are typically used
  Other Names: Extrinsic vital bleaching
  Arms: Tooth Whitening Incentive
Behavioral: Motivational Counseling — Normally three counseling sessions. Session #1: Introductions; discuss habits, feelings, pros and cons of smoking; degree of addiction; previous quit attempts and relapse; reinforce patient confidence; open-ended questions to illicit self-efficacy; homework includes Pack-Track and Why Test. Session #2: Discuss smoking patterns, triggers, and risk situations; discuss methods to resist triggers, need for medications; prepare environment and back-up plan; discuss quit date; homework to review self-help workbook. Session #3: Reinforce previous concepts; review resistance plan; discuss and arrange pharmaceutical cessation aids; set quit date; homework to finalize all self/home preparations; offer tooth polishing on quit date; follow-up by telephone or appointment.
  Other Names: Motivational Interviewing

SUMMARY:
The objectives of this study are:

1. To determine the effect that an intensive, community dental clinic centered, stop-smoking program using a motivational interviewing approach has upon cessation rates for interested, smoking inner-city dental patients.
2. To determine the effect that providing a tooth whitening incentive, in a community dental clinic stop-smoking program, has upon cessation rates for interested, smoking inner-city dental patients.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* current smoker
* dental clinic patient
* interested in quitting smoking

Exclusion Criteria:

* minors
* those unable to provide own consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | 1-year
  1-year abstinence from tobacco use, biochemically verified by carbon monoxide breath test

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Brothwell, DMD MSc, Principal Investigator — University of Manitoba
Locations (1):
- Access Downtown Dental Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided